CLINICAL TRIAL: NCT04547322
Title: The Effect of Virtual Reality on Preoperative Anxiety in Patients Undergoing Colorectal Surgery
Brief Title: Effect of Virtual Reality on Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulay ALTUN UGRAS, Associate Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gulay Ugras
Record Dates: First submitted 2020-08-26; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Preoperative Anxiety
Keywords: colorectal surgery; virtual reality; nurse

STUDY DESIGN:
Intervention Model Description: prospective, parallel, two arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: The researchers involved in the data analysis and statistics stages were blinded to the group assignment, too. However, those involved in the running of the study were not blinded. Also, the person who performed the measurements was not blinded due to the nature of VR application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR application group (Experimental): The experimental group received VR application in the preoperative period for 10 minutes.
  Interventions: Other: VR application group
- Control group (No Intervention): The control group received the routine procedure in the unit clinic where the study was conducted. The routine procedure of the unit includes patients are taken to the operating room on a stretcher and wait on the stretcher in the surgery waiting room until the operation room is prepared.

INTERVENTIONS:
Other: VR application group — During the transfer from the general surgery clinic to the operating room (3-5 minutes) and in the surgery waiting room, the VR aplication group were asked to wear a virtual reality headset (VR BOX 2) and headphones minimizing sound loss (Earpods with Apple Lightning Connector) that are compatible with mobile phones with IOS operating system. The VR headset and the headphones were controlled by a mobile phone (iPhone 7 Plus). The researchers had the patients watch three-dimensional videos (e.g. underwater world, museum trips, forest and park walks, beach trips, and space travel) for 10 minutes with their preferred background and relaxing music.
  Arms: VR application group

SUMMARY:
The aim of this study was to determine the effect of virtual reality (VR) on the preoperative anxietyof patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
The sample of this study consisted of 86 patients in experimental and control groups. The experimental group received VR application in the preoperative period for 10 minutes. Anxiety level was assessed with the Anxiety Specific to Surgery Questionnaire (ASSQ) and measured with physiological responses of anxiety such as systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), respiratory rate (RR) and peripheral oxygen saturation (SpO2) before and after VR application.

ELIGIBILITY:
Inclusion Criteria:The study included

* conscious,
* orientated and cooperated patients who could speak and understand Turkish,
* who had no psychiatric diseases,
* who were 18 years old and older,
* who were scheduled for elective colorectal surgery for the first time,
* who did not take any sedative drugs before surgery, and
* who gave written and oral permission to participate in the study

Exclusion Criteria:n The study excluded

* had language problems,
* underwent emergency surgery,
* were over 65 years of age and
* refused to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change Anxiety Specific to Surgery Questionnaire score | 10 minute
  The psychological response of patients to preoperative anxiety was evaluated with Anxiety Specific to Surgery Questionnaire. With a total of 10 items, responses are made on a five-point Likert scale format ranging from 1 (do not agree at all) to 5 (completely agree). Anxiety Specific to Surgery Questionnaire score is obtained by adding the answers to all items (minimum score=10; maximum score=50). The increase in the scale score indicates that the level of anxiety increases.
  The researchers administered Anxiety Specific to Surgery Questionnaire to all the patients before their transfer from the general surgery unit to the operating room, to the experimental group after virtual reality application, and to the control group 10 minutes after the first measurement.

SECONDARY OUTCOMES:
Change systolic blood pressure | 10 minute
  Determine patients' physiological responses (systolic blood pressure) of preoperative anxiety after virtual reality application
  The researchers measured systolic blood pressure to all the patients before their transfer from the general surgery unit to the operating room, to the experimental group after virtual reality application, and to the control group 10 minutes after the first measurement. At the same time, their systolic blood pressure values were followed on the portable monitor (Vismo, Nihon Kohden, Germany).
Change diastolic blood pressure | 10 minute
  Determine patients' physiological responses (diastolic blood pressure) of preoperative anxiety after virtual reality application
  The researchers measured diastolic blood pressure to all the patients before their transfer from the general surgery unit to the operating room, to the experimental group after virtual reality application, and to the control group 10 minutes after the first measurement. At the same time, their diastolic blood pressure values were followed on the portable monitor (Vismo, Nihon Kohden, Germany)
Change heart rate | 10 minute
  Determine patients' physiological responses (heart rate) of preoperative anxiety after virtual reality application
  The researchers measured heart rate to all the patients before their transfer from the general surgery unit to the operating room, to the experimental group after virtual reality application, and to the control group 10 minutes after the first measurement. At the same time, their heart rate were followed on the portable monitor (Vismo, Nihon Kohden, Germany)
Change respiratory rate | 10 minute
  Determine patients' physiological responses (respiratory rate) of preoperative anxiety after virtual reality application
  The researchers measured respiratory rate to all the patients before their transfer from the general surgery unit to the operating room, to the experimental group after virtual reality application, and to the control group 10 minutes after the first measurement. At the same time, their respiratory rate were followed on the portable monitor (Vismo, Nihon Kohden, Germany)
Change peripheral oxygen saturation | 10 minute
  Determine patients' physiological responses ( peripheral oxygen saturation) of preoperative anxiety after virtual reality application
  The researchers measured peripheral oxygen saturation to all the patients before their transfer from the general surgery unit to the operating room, to the experimental group after virtual reality application, and to the control group 10 minutes after the first measurement. At the same time, their peripheral oxygen saturation were followed on the portable monitor (Vismo, Nihon Kohden, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Altun Ugras, PhD, Principal Investigator — Mersin University, Nursing Faculty
Locations (1):
- Mersin University Hospital, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No